CLINICAL TRIAL: NCT01347775
Title: Inspiratory Muscle Training in Patients With End Stage Renal Failure: a Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training in Patients With End Stage Renal Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Queensland (Other)
Responsible Party: Dr Jennifer Paratz, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMTRF-06001
Record Dates: First submitted 2011-04-29; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Renal Failure; Chronic Renal Insufficiency
Keywords: Renal failure; Respiratory muscles; Resistance training
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham inspiratory muscle training (Sham Comparator): Patients in the sham group used the threshold trainer (Threshold at IMT device URES HS730, Respironics, New Jersey, Inc, Cedar Grove, NJ, USA), with the diaphragm removed.
  Interventions: Device: Sham inspiratory muscle training (URES HS730)
- Inspiratory muscle training (Experimental): Inspiratory muscle training will be by a threshold trainer (Threshold at IMT device URES HS730, Respironics, New Jersey, Inc, Cedar Grove, NJ, USA), a commercially available spring-loaded inspiratory muscle training device. It will be set at 40% of the subjects baseline maximal inspiratory pressure and increased by 10% each week by an unblinded assistant. All subjects were trained with these devices for 8-10 breaths, 3 times a day, everyday for 6 weeks
  Interventions: Device: Inspiratory muscle training (URES HS730)

INTERVENTIONS:
Device: Inspiratory muscle training (URES HS730) — It will be set at 40% of the subjects baseline maximal inspiratory pressure and increased by 10% each week by an unblinded assistant. All subjects were trained with these devices for 8-10 breaths, 3 times a day, everyday for 6 weeks
  Other Names: Threshold at IMT device URES HS730, Respironics
  Arms: Inspiratory muscle training
Device: Sham inspiratory muscle training (URES HS730) — Subjects in the control group underwent sham training, using the same device with the diaphragm removed, thus providing no resistance. They were not given frequency or duration but told to use the device when desired.
  Other Names: Threshold at IMT device URES HS730, Respironics
  Arms: Sham inspiratory muscle training

SUMMARY:
This study will investigate whether inspiratory muscle training in patients with end stage renal failure can improve strength and function.

DETAILED DESCRIPTION:
Patients with chronic renal failure commonly have weak respiratory muscles leading to problems in everyday activities and respiratory infections.

This project aims to investigate if threshold inspiratory muscle training improves the strength, everyday function and participation of patients on haemodialysis. Forty eight patients will be recruited in a randomized controlled trial of inspiratory muscle training vs sham training.

Outcome measures include the maximal inspiratory pressure and the Frenchay activities index. Initial data will be collected by a blinded assessor; the patients will train at 40 % of initial maximal inspiratory pressure for six weeks and be reassessed. If the inspiratory muscle training is effective, it will improve both the physical and functional components of the patient's lives and be recommended for all renal patients.

ELIGIBILITY:
Inclusion Criteria:

* documented chronic renal failure
* attending either haemodialysis or pre-dialysis clinic
* age 18
* English speaking
* no prior experience with inspiratory training devices.

Exclusion Criteria:

* lung collagen disorders
* renal diseases associated with autoimmune pulmonary diseases
* current pleural effusion
* pulmonary oedema
* decreased conscious level
* behavioural disturbances
* unable or refused to give consent
* taking medications that influence respiratory muscle function (e.g. steroids or cyclophosphamide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | Change between baseline (enrolment) and 6 weeks
  American Thoracic Society standards

SECONDARY OUTCOMES:
Frenchay activities index | Change between baseline (enrolment) and 6 weeks
  The Frenchay activities index is a measure of instrumental activities of everyday living.The FAI assesses a broad range of activities associated with everyday life including social and family participation

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Paratz, PhD, Principal Investigator — The University of Queensland
Locations (1):
- Royal Brisbane & Womens Hospital, Brisbane, Queensland, Australia